CLINICAL TRIAL: NCT02794636
Title: Analysis of the Clinical and Economic Impact of Adverse Events and Medication-related Toxicities Associated With Interferon (IFN) Treatment for Patients With Stage III Melanoma
Brief Title: Interferon Toxicities in Melanoma Treatment
Acronym: ITMT
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA184-404
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Stage III Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IFN Treatment: Adult (age ≥ 18 years) patients identified as having stage III melanoma and no other primary or secondary cancer who initiated treatment with IFN between 1/1/2007 and 12/31/2011. Patients are required to have continuous pharmaceutical benefit enrollment for 180 days before (pre-index) and after (post-index) IFN initiation and no evidence of treatment with systemic chemotherapy during the pre- or post-index period

SUMMARY:
The primary objective of this study is to quantify and compare the prevalence of adverse events (AEs) in patients with stage III melanoma before and after initiation of interferon (IFN) therapy in a real-world setting. A secondary objective is to quantify annual costs and resource utilization before and after IFN initiation among patients with stage III melanoma in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pharmacy claim for IFN between 1/1/2007 and 12/31/2011. The date of the first observed claim will be defined as the index date
* Patients with a melanoma diagnosis based on two medical claims prior to the index date
* Patients with a procedure code for melanoma-related lymph node dissection before the index date
* Patients ≥ 18 years of age on or before the index date
* Patients with continuous benefit enrollment for at least 180 days before and after the index date

Exclusion Criteria:

* Patients with diagnosis of any other (primary) cancer during the 180-day pre-index period (excepting skin cancers and hematologic malignancies)
* Patients with diagnosis of a secondary cancer during the 180-day pre-index period or on the index date (excepting lymph node metastasis to a site common for melanoma or an improbable site for any other primary cancer)
* Patients who received systemic chemotherapy during the pre- or post-index period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Health plan enrollees whose data are reflected in the Truven Health MarketScan Commercial and Medicare Supplemental database. This database captures clinical utilization, expenditures and enrollment across inpatient, outpatient, prescription drug, and carve-out services from a selection of large employers, health plans, and government and public organizations
Sampling Method: Non-Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of depression in patients with stage III melanoma before initiation of Interferon alfa-2b (IFN) therapy | 180 days prior to the index date
Prevalence of depression in patients with stage III melanoma after initiation of IFN therapy | 180 days after the index date
Prevalence of fatigue in patients with stage III melanoma before initiation of IFN therapy | 180 days prior to the index date
Prevalence of fatigue in patients with stage III melanoma after initiation of IFN therapy | 180 days after the index date
Prevalence of myalgia in patients with stage III melanoma before initiation of IFN therapy | 180 days prior to the index date
Prevalence of myalgia in patients with stage III melanoma after initiation of IFN therapy | 180 days after the index date

SECONDARY OUTCOMES:
Pre-IFN treatment period Health care costs related to depression | 180 days prior to the index date
Post-IFN treatment period Health care costs related to depression | 180 days after the index date
Pre-IFN treatment period Health care costs related to fatigue | 180 days prior to the index date
Post-IFN treatment period Health care costs related to fatigue | 180 days after the index date
Pre-IFN treatment period Health care costs related to myalgia | 180 days prior to the index date
Post-IFN treatment period Health care costs related to myalgia | 180 days after the index date

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx